CLINICAL TRIAL: NCT02884583
Title: Association Between Asthma and Food Allergy in Children and Adults
Brief Title: Association Between Asthma and Food Allergy
Acronym: AAAli
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9613
Record Dates: First submitted 2016-07-18; First posted 2016-08-31 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2016-08

CONDITIONS: Food Allergy Suspected; Food Allergy Proved
Keywords: Food allergy; asthma; Predictive factor; Exacerbation; Prevalence
MeSH Terms: conditions — Food Hypersensitivity; Asthma | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pulmonary function test (Experimental): Patients hospitalized for Oral Food Challenge realize pulmonary function test
  Interventions: Other: Pulmonary function test

INTERVENTIONS:
Other: Pulmonary function test — Patients hospitalized for OFC realise a Resting pulmonary function tests (PFT) which include the assessment of ventilatory capacity: spirometry (forced expiratory flows and mobilisable volumes) and static volume assessment, by using body plethysmography, were realized before, during and after the OFC. An exhaled fraction of NO (FeNO) is also realized to characterize asthma.

SUMMARY:
Prevalences of food allergies and asthma increased in the population during the last decades. These two pathologies, responsible for a real burden, are often associated and are to be considered as comorbidities; this aspect is more and more studied in the literature and many authors tried to find a link between diets and asthma. The narrow link between these two atopic pathologies and the fact that food allergy can come along with respiratory symptoms also in patients without history of asthma must be better understood, considered into the management of food allergy. The main objective of this study is to study the prevalence of signs and/or symptoms suggestive of bronchial hyperreactivity, during an oral food challenge (OFC) in patients older than 5 years. The secondary objective is to study the risk factors to develop asthma during a food allergy reaction.

This historical-prospective single center study , was realized in the Allergy Unit of the University Hospital of Montpellier. All the patients having been hospitalized for a positive OFC between January, 2001 and January, 2016 were included. The diagnosis of asthma was established according to the recommended international clinical and physiological criteria. Prevalence of bronchial hyperreactivity during OFC among those with positive OFC, was calculated. The search for risk factors was made by a logistic regression univariate then multivariate, completed by a decision tree.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized for oral food challenge at the hospital

Exclusion Criteria:

* Patient want to leave the protocol
* Patient take medication forbidden during the study

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-04-26 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Number of patient with bronchospasm in OFC | up to 3 hours

SECONDARY OUTCOMES:
Questionnaire for the assessment of the responsible food of allergy | up to 3 hours
the eliciting dose | up to 3 hours
  the dose of the tested food which elicits the symptoms of allergy
The grade of the allergic reaction shown during the last food ingestion of the concerned food | up to 3 hours
The presence of one or several sensitisations associated with respiratory allergens | up to 3 hours
  defining the atopic ground
The level of specific immunoglobulin E of the concerned food | up to 3 hours
The time of appearance of the first signs of atopy | up to 3 hours
questionnaire for the assessment of the mode of clinical expression of food allergies | up to 3 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided